CLINICAL TRIAL: NCT01526317
Title: A Randomized, Open Label, Cross-over Clinical Trial to Investigate Pharmacokinetics and Drug Interaction of Crestor and Glucodown OR SR in Healthy Volunteers
Brief Title: A Phase 1 Clinical Trial to Investigate Pharmacokinetics and Drug Interaction of Crestor and Glucodown OR SR in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YH14755-101
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Pharmacokinetics and Drug Interaction of Crestor and Glucodown SR
Keywords: Drug interaction; Rosuvastatin; Metformin SR; Pharmacokinetic
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): This arm is consist of 6 subject. Crestor 10mg and Glucodown 750mg for 5 day during period 1. Crestor 10mg alone for 5 day during period 2. Glucodown 750mg alone for 5 day during period 3.
  Interventions: Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg)
- 2 (Experimental): This arm is consist of 6 subject. Glucodown 750mg alone for 5 day during period 1. Crestor 10mg and Glucodown 750mg for 5 day during period 2. Crestor 10mg alone for 5 day during period 3.
  Interventions: Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg)
- 3 (Experimental): This arm is consist of 6 subject. Crestor 10mg alone for 5 day during period 1. Glucodown 750mg alone for 5 day during period 2. Crestor 10mg and Glucodown 750mg for 5 day during period 3.
  Interventions: Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg)
- 4 (Experimental): This arm is consist of 6 subject. Glucodown 750mg alone for 5 day during period 1. Crestor 10mg alone for 5 day during period 2. Crestor 10mg and Glucodown 750mg for 5 day during period 3.
  Interventions: Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg)
- 5 (Experimental): This arm is consist of 6 subject. Crestor 10mg alone for 5 day during period 1. Crestor 10mg and Glucodown 750mg for 5 day during period 2. Glucodown 750mg alone for 5 day during period 3.
  Interventions: Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg)
- 6 (Experimental): This arm is consist of 6 subject. Crestor 10mg and Glucodown 750mg for 5 day during period 1. Glucodown 750mg alone for 5 day during period 2. Crestor 10mg alone for 5 day during period 3.
  Interventions: Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg)

INTERVENTIONS:
Drug: Crestor 10mg(Rosuvastatin 10mg), Glucodown OR SR 750mg(Metformin SR 750mg) — For co-administration,Crestor 1 tablet and Glucodown 1 tablet a day for 5 day.(1 period) For separate administration, Crestor 1 tablet a day for 5 day and Glucodown 1 tablet a day for 5 day.

SUMMARY:
This clinical trial is designed to compare the pharmacokinetic characteristics of combination and separate administration of Crestor(Rosuvastatin) and Glucodown(Metformin SR). Also investigate drug interaction between separate and combination administration.

Total number of subjects is 36. 6 group(6 for 1 group), 3 period, consecutive 5 day administration, 10 days washout after 5th day of administration.

All subjects take Crestor alone, Glucodown alone, Crestor+Glucodown combination during 3 each period.

ELIGIBILITY:
Inclusion Criteria:

* 20~50 yrs old, healthy Korean Subjects
* Body weight <ideal body weight±20%
* No congenital, chronic disease, No current disease
* Subjects who are diagnosed to include by medical doctor from laboratory and ECG result.
* Subjects who agree to keep contraceptive methods during the clinical trial.

Exclusion Criteria:

* Subjects who are allergic to investigational drug.
* Subjects who have a medical history which can affect the clinical trial.
* Hypertension(Systolic BP ≥ 150mmHG or Diastolic BP ≥ 100mmHg), Hypotension(Systolic BP ≤ 100mmHg or Diastolic BP ≤ 65mmHg)
* Subjects who have taken other medicine in recent 2~4 weeks.
* Subjects who have a risk of hypoglycemia and imbalance in taking a diet.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
AUCtau | 72 hr
Css,max | 72 hr

SECONDARY OUTCOMES:
AUCss,last | 72 hr
AUCss,inf | 72 hr
Css,min | 72 hr
Tss,max | 72 hr
t1/2 | 72 hr

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsu Park, MD, Ph.D, Principal Investigator — Severance Hospital, Yonsei University
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Lee D, Roh H, Son H, Jang SB, Lee S, Nam SY, Park K. Pharmacokinetic interaction between rosuvastatin and metformin in healthy Korean male volunteers: a randomized, open-label, 3-period, crossover, multiple-dose study. Clin Ther. 2014 Aug 1;36(8):1171-81. doi: 10.1016/j.clinthera.2014.06.004. Epub 2014 Jun 26. PMID 24976448